CLINICAL TRIAL: NCT03006809
Title: Optimal Fecal Microbiota Transplant Dosing for Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Najwa Elnachef (Other)
Responsible Party: Sponsor-Investigator, Najwa Elnachef, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-20066
Record Dates: First submitted 2016-12-21; First posted 2016-12-30 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; FMT; fecal transplant
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Vancomycin; Metronidazole; Neomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): pretreatment antibiotics + FMT delivered by colonoscopy + FMT capsules per week x 6 weeks
  Interventions: Biological: Fecal Microbiota Transplantation (FMT), OpenBiome; Other: pretreatment antibiotics
- 2 (Experimental): no antibiotics, FMT delivered by colonoscopy + FMT capsules per week x 6 weeks
  Interventions: Biological: Fecal Microbiota Transplantation (FMT), OpenBiome
- 3 (Experimental): pretreatment antibiotics + FMT delivered by colonoscopy + FMT delivered by enema once per week x 6 weeks
  Interventions: Biological: Fecal Microbiota Transplantation (FMT), OpenBiome; Other: pretreatment antibiotics
- 4 (Experimental): no antibiotics, FMT delivered by colonoscopy + FMT delivered by enema once per week x 6 weeks
  Interventions: Biological: Fecal Microbiota Transplantation (FMT), OpenBiome

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT), OpenBiome — Delivered by colonoscopy, enema or orally (as capsules)
Other: pretreatment antibiotics — 5 day course (vancomycin PO 500mg bid, metronidazole PO 500mg bid, and neomycin PO 500mg bid) starting 6 days prior FMT
  Other Names: vancomycin, metronidazole, neomycin
  Arms: 1; 3

SUMMARY:
This is a prospective unblinded, randomized trial for the use of Fecal Microbiota Transplantation (FMT) for the treatment of Ulcerative Colitis (UC), in combination with or without antibiotic pretreatment.

DETAILED DESCRIPTION:
This is a prospective open-label, randomized trial for the use of Fecal Microbiota Transplantation (FMT) for the treatment of Ulcerative Colitis (UC), in combination with or without antibiotic pretreatment.

This trial involves 11 study visits at UCSF in San Francisco, CA.

The routes of administration will be via colonoscopy for all subjects with maintenance therapy administered orally (i.e. using encapsulated FMT) for half of the subjects and per rectum by enema in the other half of the subjects. Additionally, the utility of pretreatment antibiotics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of mild to moderate Ulcerative Colitis confirmed by endoscopy and pathology.
* Total Mayo score 4-9, endoscopic subscore ≥1; patients who have not had endoscopic evaluation within one year of enrollment will have flexible sigmoidoscopy for evaluation.
* Age 18 - 64 and deemed otherwise healthy at the discretion of the investigator.
* Concurrent therapies with mesalamine (stable x 4 weeks), immunomodulators (stable x 3 months), and biologic agents (stable x 3 months) will be allowed to continue during study.
* If patient is on prednisone, the dose must be ≤ 10mg/day at the time of treatment and will be weaned by 2.5mg/week during the study period.

Exclusion Criteria:

* Severe or refractory UC defined as Mayo score ≥10, endoscopic disease activity score 3
* Untreated enteric infection (positive stool test for any of the following: Clostridium difficile, Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic E. coli or other enteric infection at the discretion of the investigator.
* History of colectomy
* Disease limited to distal proctitis
* Patients taking probiotics within 6 weeks of planned FMT therapy.
* Severe immunodeficiency, inherited or acquired (e.g. HIV, chemotherapy or radiation therapy)
* Patients with the following laboratory abnormalities: absolute neutrophil count (ANC) < 1000 / µl, platelets <50 x 10^9 /L,, hemoglobin <6.5 g/dL..
* History of anaphylaxis (severe allergic reaction) to food allergens (e.g. tree nuts, shellfish)
* Dysphagia (oropharyngeal, esophageal, functional, neuromuscular)
* History of recurrent aspiration episodes
* Documented severe gastroparesis
* Active intestinal obstruction
* Patients with renal insufficiency (GFR < 50ml/min)
* Allergy to the following generally regarded as safe ingredients (GRAS): glycerol, acid resistant HPMC, gellan gum, cocoa butter, titanium dioxide
* Adverse event attributable to any previous FMT
* Allergy/intolerance to proton pump inhibitor therapy
* Allergy/intolerance to vancomycin, metronidazole, or neomycin.
* Non-steroidal inflammatory medications (NSAIDs) as long-term treatment, defined as use for at least 4 days a week each month.
* Cholestyramine use
* Any condition in which the investigator thinks the FMT treatment may pose a health risk (e.g. severely immunocompromised)
* Simultaneous participation in another interventional clinical trial
* Patients who are pregnant, breast feeding or planning pregnancy during study trial period.
* During the trial period until one week after the trial end: Non-use of appropriate contraceptives in females of childbearing potential (e.g. condoms, intrauterine device (IUD), hormonal contraception, or other means considered adequate by the responsible investigator) or in males with a child-fathering potential (condoms, or other means considered adequate by the responsible investigator during treatment) or well-founded doubt about the patient's cooperation
* Patients with any other significant medical condition that could confound or interfere with evaluation of safety, tolerability or prevent compliance with the study protocol at the discretion of the investigator
* Life expectancy <6 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
The occurrence of a Serious Adverse event (SAE), solicited and unsolicited AE, new gastrointestinal medical condition and diagnoses from FMT treatment or new infection from FMT treatment | up to 1 year
  safety endpoint
Steroid-free Clinical Remission at week 9 + endoscopic remission or response defined as total Mayo score ≤ 2 with all four sub-scores ≤ 1 and a ≥ 1 point reduction in endoscopy sub-score | 8 weeks post initial treatment

SECONDARY OUTCOMES:
Changes in microbiome with FMT therapy. Changes in the microbiome: assessed by frequent stool sampling for 16S rRNA analysis prior to each FMT therapy and after the last capsule/enema dose | up to 1 year
Clinical Response: decrease in Mayo score by ≥ 3 points, decrease in bleeding subscore by ≥ 1, or absolute subscore of 0-1 | 8 weeks post initial treatment
Progression of disease defined by initiation of anti-TNF agents or Corticosteroids: Initiation of anti-TNF agents (such as infliximab, adalimumab, certolizumab, vedolizumab and steroids). Includes time gap until additional agents are started. | 2, 4 and 8 weeks post initial FMT
Progression of disease defined by increase in dosages of current UC medications | 2, 4 and 8 weeks post initial FMT
Progression of disease defined by time to colectomy | up to one year post initial FMT
Time to death secondary to UC | up to one year post initial FMT
Progression of disease defined by clinical flare (Time to next flare) | 2, 4 and 8 weeks post initial FMT
Increase in Quality of Life (based on RAND SF-36 survey and score) | 8 weeks post initial FMT
Changes in Mood/Depression Score (based on PHQ-9 survey and score) | 8 weeks post initial FMT

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Division of Gastroenterology at Mount Zion, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith BJ, Piceno Y, Zydek M, Zhang B, Syriani LA, Terdiman JP, Kassam Z, Ma A, Lynch SV, Pollard KS, El-Nachef N. Strain-resolved analysis in a randomized trial of antibiotic pretreatment and maintenance dose delivery mode with fecal microbiota transplant for ulcerative colitis. Sci Rep. 2022 Apr 1;12(1):5517. doi: 10.1038/s41598-022-09307-5. PMID 35365713